CLINICAL TRIAL: NCT07022158
Title: Relationship Between Antenatal Body Shape Index and Pregnancy Complications
Brief Title: Antenatal Body Shape Index and Pregnancy Complications
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Elif Betul Esmer, Principal Investigator, Obstetrics and Gynaecology Specialist, Abant Izzet Baysal University
Other Study IDs: AbantIBU-elifbetulesmer-001
Record Dates: First submitted 2025-05-23; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Gestational Complications; Body Mass Index; Waist Circumference; Gestational Hypertension; Gestational Diabetes Mellitus (GDM); Preeclampsia (PE)
Keywords: gestational hypertension; gestational diabetes; preeclampsia; body shape index; waist circumference
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Diabetes, Gestational; Pre-Eclampsia | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 184 pregnant women who applied to Bolu Abant İzzet Baysal Training and Research Hospital
  Interventions: Other: The patients participating in the study were between 6 and 16 weeks of pregnancy. Height, body weight, and waist circumference were measured at the first antenatal visit at 2 weeks.

INTERVENTIONS:
Other: The patients participating in the study were between 6 and 16 weeks of pregnancy. Height, body weight, and waist circumference were measured at the first antenatal visit at 2 weeks. — 170 patients at 6-16th weeks of gestation were prospectively analyzed. Body mass index (BMI) and ABSI were calculated. Patients were analyzed according to the presence of GDM, GHT and preeclampsia at follow-up.

SUMMARY:
Background/aim: Gestational diabetes (GDM), gestational hypertension (GHT) and preeclampsia are common complications of pregnancy. In this study, it was aimed to determine the relationship between body shape index (ABSI), calculated based on antenatal measurements of the height, weight and waist circumference, and GDM, GHT and preeclampsia.

Materials and methods: 170 patients at 6-16th weeks of gestation were prospectively analyzed. Body mass index (BMI) and ABSI were calculated. Patients were analyzed according to the presence of GDM, GHT and preeclampsia at follow-up.

Our study is the first in terms of its subject and makes a significant contribution to the literature.

ELIGIBILITY:
Inclusion Criteria:

* Having a singleton pregnancy
* Pregnancy follow-up and birth must have taken place at Bolu Abant İzzet Baysal University Training and Research Hospital.
* Voluntary informed consent form must be signed to participate in the study.

Exclusion Criteria:

* Multiple pregnancies
* Additional systemic and chronic diseases (chronic hypertension, DM, hepatic diseases such as cholestasis, cardiac diseases, rheumatic diseases, renal diseases…)
* History of Gestational Diabetes, Gestational Hypertension and Preeclampsia in previous pregnancies

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 170 patients at 6-16th weeks of gestation
Sampling Method: Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Calculation of body shape index at 6-16 weeks of gestation | 6-16 weeks of gestation
  The study included pregnant women who applied to the Obstetrics and Gynecology outpatient clinic of Bolu Abant İzzet Baysal Training and Research Hospital between September 2023 and March 2024. During the first antenatal examination of the patients at 6-16 weeks of pregnancy, body shape indexes were calculated by measuring height, body weight and waist circumference.

SECONDARY OUTCOMES:
Number of patients developing pregnancy complications | gestation period and first 6 weeks postpartum
  Patients whose body shape index was calculated at 6-16 weeks of gestation were evaluated during pregnancy follow-up according to the development of Gestational Diabetes, Gestational Hypertension and Preeclampsia.

CONTACTS AND LOCATIONS:
Locations (1):
- Abant Izzet Baysal University Faculty of Medicine, 14030, Bolu, Turkey, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No